CLINICAL TRIAL: NCT02177136
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose-Finding, Clinical Trial Evaluating the Efficacy and Safety of Obeticholic Acid in Subjects With Primary Sclerosing Cholangitis
Brief Title: Obeticholic Acid (OCA) in Primary Sclerosing Cholangitis (PSC)
Acronym: AESOP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intercept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 747-207; 2014-002205-38 (EudraCT Number)
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Results first posted 2018-05-30 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Primary Sclerosing Cholangitis (PSC)
Keywords: PSC
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — obeticholic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Following completion of the DB phase, participants were asked to reconfirm their consent for participation in the open-label LTSE phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1.5 mg OCA titrating to 3 mg OCA (Experimental): Participants randomized to 1.5 mg OCA took 1.5 mg OCA daily for 12 weeks during the DB phase. If tolerated, the dose was increased to 3 mg OCA daily for an additional 12 weeks.
  Interventions: Drug: Obeticholic Acid (OCA)
- 5 mg OCA titrating to 10 mg OCA (Experimental): Participants randomized to 5 mg OCA took 5 mg OCA daily for 12 weeks during the DB phase. If tolerated, the dose was increased to 10 mg OCA daily for an additional 12 weeks.
  Interventions: Drug: Obeticholic Acid (OCA)
- Placebo (Experimental): Participants randomized to placebo took placebo for 24 weeks during the DB phase.
  Interventions: Drug: Placebo
- LTSE OCA Total (Experimental): Following completion of the DB phase, participants were asked to reconfirm their consent for participation in the LTSE phase (planned as a further 24 months) beginning at 5 or 10 mg OCA, based on the last treatment received during the DB phase. Doses up to 10 mg daily were evaluated. All participants received open-label OCA during the LTSE phase of the study.
  Interventions: Drug: Obeticholic Acid (OCA)

INTERVENTIONS:
Drug: Obeticholic Acid (OCA)
  Other Names: 6alpha-ethylchenodeoxycholic acid (6-ECDCA); INT-747
  Arms: 1.5 mg OCA titrating to 3 mg OCA; 5 mg OCA titrating to 10 mg OCA; LTSE OCA Total
Drug: Placebo
  Arms: Placebo

SUMMARY:
This was a phase 2, double-blind (DB), placebo-controlled trial in participants with primary sclerosing cholangitis to evaluate the effect of obeticholic acid on liver biochemistry, in particular, serum alkaline phosphatase; and, safety. The long-term safety extension (LTSE) phase was conducted to evaluate the safety, tolerability, and efficacy of long-term, open-label use of OCA in participants with PSC who had completed the DB phase of the study.

DETAILED DESCRIPTION:
This was a phase 2, randomized, double-blind, placebo-controlled, dose-finding evaluation of the efficacy and safety of OCA in participants with PSC. Approximately 75 participants who provided written informed consent and met all of the inclusion and none of the exclusion criteria were randomized to 1 of 3 treatment groups as follows: 1.5 milligrams (mg) titrating to 3 mg OCA, 5 mg titrating to 10 mg OCA, or placebo, in a 1:1:1 ratio. Participants self-administered investigational product (IP) orally, once daily for 2 consecutive 12-week periods.

For the first 12 weeks, the participant's dose was 1.5 mg OCA, 5 mg OCA, or placebo. After 12 weeks, the participant's dose was titrated as follows, providing there were no limiting safety or tolerability concerns in the opinion of the Investigator, while maintaining the trial blind: the 1.5 mg OCA treatment group titrated to 3 mg, the 5 mg OCA treatment group titrated to 10 mg OCA, and the placebo group remained on placebo. Double-blind treatment continued for a further 12 weeks at that dose.

Any participant whose dose was not titrated, due to safety or tolerability concerns, remained on their starting treatment (1.5 mg OCA, 5 mg OCA, or placebo) for the remainder of the DB phase to Week 24.

Randomization was stratified by the presence or absence of concomitant ursodeoxycholic acid (UDCA) use and total bilirubin level (≤1.5x upper limit of normal [ULN] or >1.5x ULN but <2.5x ULN).

Following completion of the DB phase, participants were asked to reconfirm their consent for participation in the open-label LTSE phase (planned as a further 24 months).

ELIGIBILITY:
Inclusion Criteria:

* Must have had a diagnosis of PSC (based on cholangiography at any point in time).
* Alkaline phosphatase at Screening ≥2x ULN.
* Total bilirubin at Screening <2.5x ULN.
* For participants with concomitant inflammatory bowel disease (IBD):

  1. Colonoscopy (if participant has a colon) or other appropriate endoscopic procedure within 12 months of Day 0 confirming no dysplasia or colorectal cancer
  2. Participants with Crohn's Disease (CD) must have been in remission as defined by a Crohn's Disease Activity Index (CDAI) <150
  3. Participants with ulcerative colitis (UC) must either have been in remission or have had mild disease. Remission was defined as a partial Mayo score of ≤2 with no individual sub-score exceeding 1. Mild disease was defined as a partial Mayo score ≤3 with no individual sub-score exceeding 1 point.
* For participants being administered UDCA as part of their standard of care, the dose must have been stable for ≥3 months prior to, and including, Day 0 and must not have exceeded 20 mg/kilograms/day during this time.
* Participants being administered biologic treatments (for example, anti-tumor necrosis factor or anti-integrin monoclonal antibodies), immunosuppressants, systemic corticosteroids, or statins, must have been on a stable dose for ≥3 months prior to, and including, Day 0 and should plan to remain on a stable dose throughout the trial.
* Contraception: female participants of childbearing potential must have used ≥1 effective method (≤1% failure rate) of contraception during the trial and until 4 weeks following the last dose of IP (including LTSE doses).

Exclusion Criteria:

* Evidence of a secondary cause of sclerosing cholangitis at Screening.
* Immunoglobulin G4 (IgG4) >4x ULN at Screening or evidence of IgG4 sclerosing cholangitis.
* Small duct cholangitis in the absence of large duct disease.
* Presence of clinical complications of chronic liver disease or clinically significant hepatic decompensation, including:

  * Current Child Pugh classification B or C
  * History of, or current diagnosis or suspicion of, cholangiocarcinoma or other hepatobiliary malignancy, or biliary tract dysplasia.
  * History of liver transplantation, or current model of end stage liver disease score ≥12
  * History of, or current, cirrhosis with complications, including history or presence of spontaneous bacterial peritonitis hepatocellular carcinoma or hepatic encephalopathy (as assessed by the Investigator)
  * Current known portal hypertension with complications, including known gastric or large esophageal varices, poorly controlled or diuretic resistant ascites, history of variceal bleeds, or related therapeutic or prophylactic interventions (for example, beta blockers, insertion of variceal bands or transjugular intrahepatic portosystemic shunt).
  * History of, or current, hepatorenal syndrome (type I or II) or Screening serum creatinine >2 mg/deciliter (178 micromoles/liter [L]).
  * Platelet count <50 x 10^9/L.
* Current clinical evidence of dominant strictures that were considered clinically relevant in the opinion of the Investigator or current biliary stent at Screening.
* Current cholecystitis or evidence of current biliary obstruction due to gallstones. Asymptomatic gallstones that were not considered a safety risk in the opinion of the Investigator might have been acceptable, subject to discussion and agreement with the Medical Monitor.
* Colonic dysplasia within ≤5 years prior to Day 0.
* History of small bowel resection.
* History of other chronic liver diseases, including, but not limited to, primary biliary cholangitis (PBC), alcoholic liver disease, non-alcoholic fatty liver disease, autoimmune hepatitis, hepatitis B virus (unless seroconverted and no positive Hepatitis B Virus deoxyribonucleic acid), hepatitis C virus and overlap syndrome.
* Known Gilbert's syndrome or history of elevations in unconjugated (indirect) bilirubin >ULN or unconjugated (indirect) bilirubin >ULN at Screening.
* Known history of human immunodeficiency virus infection.
* Currently experiencing, or experienced within ≤3 months of Screening, pruritus requiring systemic or enteral treatment.
* Known or suspected acute cholangitis in the 3 months prior to, and including, Day 0 including cholangitis treated with antibiotics.
* Administration of antibiotics is prohibited ≤1 month of Day 0 (unless participant was on a stable prophylaxis dose for at least 3 months prior to Day 0).
* Administration of the following medications was prohibited ≤6 months of Day 0 and throughout the trial: fenofibrate or other fibrates and potentially hepatotoxic medications (including alpha-methyl-dopa, sodium valproic acid, isoniazide, or nitrofurantoin).
* IBD flare during Screening (up to and including Day 0), where "flare" was defined as follows:

  * UC flare: partial Mayo Score ≥5, and
  * CD flare: CDAI ≥250
* Evidence of deleterious effects of alcohol abuse (as assessed by the Investigator) or excessive alcohol consumption (>4 units/day for males, >2 units/day for females).
* Known or suspected use of illicit drugs or drugs of abuse (allowed if medically prescribed or indicated) within 3 months of Day 0.
* If female: known pregnancy, or had a positive urine pregnancy test (confirmed by a positive serum pregnancy test), or lactating.
* Other concomitant disease, malignancy, or condition likely to significantly decrease life expectancy to less than the duration of the trial (for example, moderate to severe congestive heart failure).
* Participation in another investigational drug, biologic, or medical device trial within 30 days prior to Screening.
* History of noncompliance with medical regimens, or participants who were considered to be potentially unreliable.
* Blood or plasma donation within 30 days prior to Day 0.
* Mental instability or incompetence such that the validity of informed consent or compliance with the trial was uncertain.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2015-02-09 (Actual); Primary Completion 2017-03-07 (Actual); Study Completion 2018-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Harb, MD, Study Chair — Intercept Pharmaceuticals, Inc.
Locations (36):
- United States (33):
  - St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - University of California Davis Medical Center, Sacramento, California
  - University of Colorado, Denver, Aurora, Colorado
  - University of Miami Hospital, Miami, Florida
  - Piedmont Atlanta Georgia Transplant Institute, Atlanta, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Tulane Medical Center, New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Southern Therapy and Advanced Research, Jackson, Mississippi
  - St. Louis University Gastroenterology & Hepatology, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - CHI St. Luke's Health Baylor College of Medicine Medical Center, Houston, Texas
  - Liver Associates of Texas, P.A., Houston, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - McGuire DVAMC, Richmond, Virginia
  - Swedish Organ Transplant and Liver Center, Seattle, Washington
- Italy (3):
  - Dipartimento di Universitario di Scienze Mediche e Chirurgiche, Bologna
  - Azienda Socio Sanitaria Territoriale di Monza, Monza
  - Azienda Ospedaliera Universita di Padova - Struttura Operativa Complessa Gastroenterologia, Padua

REFERENCES:
- [Result] Kowdley KV, Vuppalanchi R, Levy C, Floreani A, Andreone P, LaRusso NF, Shrestha R, Trotter J, Goldberg D, Rushbrook S, Hirschfield GM, Schiano T, Jin Y, Pencek R, MacConell L, Shapiro D, Bowlus CL; AESOP Study Investigators. A randomized, placebo-controlled, phase II study of obeticholic acid for primary sclerosing cholangitis. J Hepatol. 2020 Jul;73(1):94-101. doi: 10.1016/j.jhep.2020.02.033. Epub 2020 Mar 10. PMID 32165251

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started December 2014 and completed September 2016. All participants were required to undergo thorough screening procedures, to confirm they met the eligibility criteria, during the 30-day period preceding the first dose.
Pre-assignment Details: Double-blind (DB) Phase: 77 participants were randomly allocated to treatment with placebo, 1.5 milligrams (mg) obeticholic acid (OCA) titrated to 3 mg OCA, or 5 mg OCA titrated to 10 mg OCA; however, 1 participant did not receive treatment. Long-term Safety Extension (LTSE): Open-label OCA doses up to 10 mg daily were evaluated.
Groups:
- Placebo: Participants randomized to placebo took placebo daily for 24 weeks during the DB phase.
Period: DB Phase
Arm/Group | 1.5 mg OCA Titrating to 3 mg OCA | 5 mg OCA Titrating to 10 mg OCA | Placebo | LTSE OCA Total
Started | 26 | 26 | 25 | 0
Received At Least 1 Dose Of Study Drug | 25 (One participant randomized to receive 1.5 mg OCA titrating to 3 mg OCA withdrew prior to dosing.) | 26 | 25 | 0
Completed | 19 | 21 | 21 | 0
Not Completed | 7 | 5 | 4 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Discontinued Due to Pruritus | 1 | 3 | 0 | 0
Not completed — Adverse Event | 3 | 2 | 3 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Withdrew Consent Prior to Dosing | 1 | 0 | 0 | 0
Period: LTSE Phase
Arm/Group | 1.5 mg OCA Titrating to 3 mg OCA | 5 mg OCA Titrating to 10 mg OCA | Placebo | LTSE OCA Total
Started | 0 (Eligible participants who completed the DB phase could enroll in the LTSE phase.) | 0 (Eligible participants who completed the DB phase could enroll in the LTSE phase.) | 0 (Eligible participants who completed the DB phase could enroll in the LTSE phase.) | 59 (Eligible participants who completed the DB phase could enroll in the LTSE phase.)
Received At Least 1 Dose Of Study Drug (All participants received open-label OCA during the LTSE phase of the study.) | 0 | 0 | 0 | 59
Completed | 0 | 0 | 0 | 35
Not Completed | 0 | 0 | 0 | 24
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 10
Not completed — Discontinued Due to Pruritus | 0 | 0 | 0 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Participant Moved | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: A total of 77 participants were randomly allocated to treatment with placebo, 1.5 mg OCA titrated to 3 mg or 5mg OCA titrated to 10mg; however, 1 participant did not receive treatment. Therefore, the baseline analysis population of 76 participants is the Intent-to-Treat Population.
Groups:
- 1.5 mg OCA Titrating to 3 mg OCA: Participants randomized to 1.5 mg OCA took 1.5 mg OCA daily for 12 weeks. If tolerated, the dose was increased to 3 mg OCA daily for an additional 12 weeks.
- 5 mg OCA Titrating to 10 mg OCA: Participants randomized to 5 mg OCA took 5 mg OCA daily for 12 weeks. If tolerated, the dose was increased to 10 mg OCA daily for an additional 12 weeks.
- Placebo: Participants randomized to placebo took placebo for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | 1.5 mg OCA Titrating to 3 mg OCA | 5 mg OCA Titrating to 10 mg OCA | Placebo | Total
Number analyzed (Participants) | 25 | 26 | 25 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 23 | 24 | 71
  >=65 years | 1 | 3 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (12.56) | 44.9 (14.28) | 43.7 (13.05) | 43.4 (13.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 11 | 35
  Male | 15 | 12 | 14 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 5
  Not Hispanic or Latino | 23 | 24 | 24 | 71
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 3 | 10
  White | 21 | 22 | 22 | 65
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Alkaline phosphatase (ALP) [Mean (Standard Deviation); unit: units/liter (U/L)] | 422.5 (123.07) | 428.5 (178.19) | 562.8 (300.22) | 470.7 (220.20)
Total Bilirubin [Mean (Standard Deviation); unit: micromoles (umol)/L] | 16.3 (8.17) | 19.4 (10.94) | 20.9 (11.48) | 18.9 (10.35)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 74.5 (12.51) | 73.6 (12.76) | 73.0 (12.95) | 73.7 (12.59)
Height [Mean (Standard Deviation); unit: centimeter] | 174.4 (8.95) | 170.4 (11.61) | 172.6 (10.70) | 172.4 (10.49)
Body Mass Index [Mean (Standard Deviation); unit: kg/meter squared] | 24.6 (4.38) | 25.3 (3.74) | 24.5 (3.71) | 24.8 (3.92)
International Normalized Ratio (INR) [Mean (Standard Deviation); unit: ratio] — The INR is the ratio of a participant's prothrombin time to a normal (control) sample and corrected for the analytical system being used.
  ratio | 1.0 (0.06) | 1.0 (0.10) | 1.0 (0.07) | 1.0 (0.08)

OUTCOME MEASURES:

1. Primary Outcome: DB Phase: Change From Baseline In Serum Alkaline Phosphatase (ALP)
Description: The primary efficacy analysis compared the Week 24 change from Baseline in ALP between OCA treatment group and placebo using an analysis of covariance (ANCOVA) model with fixed effects for treatment group and randomization strata, and Baseline as a covariate. Results are reported in U/L.
Time Frame: Baseline, Week 24
Population: Intent-to-Treat Population: All randomized participants who received any amount of investigational product within the DB phase.
Measure: Least Squares Mean (Standard Error); unit: U/L
Groups:
- Placebo: Participants randomized to placebo took placebo daily for 24 weeks.
Arm/Group | 1.5 mg OCA Titrating to 3 mg OCA | 5 mg OCA Titrating to 10 mg OCA | Placebo
Number analyzed (Participants) | 25 | 26 | 25
U/L | -105.05 (38.02) | -110.19 (33.77) | -26.76 (36.65)
Statistical Analysis 1: Comparison: 5 mg OCA Titrating to 10 mg OCA vs Placebo; Test type: Superiority; p = 0.0434, ANCOVA; ANCOVA model with treatment group and randomization stratification factors as fixed effects and baseline as covariate
Statistical Analysis 2: Comparison: 1.5 mg OCA Titrating to 3 mg OCA vs Placebo; Test type: Superiority; p = 0.0665, ANCOVA; ANCOVA model with treatment group and randomization stratification factors as fixed effects and baseline as covariate

2. Primary Outcome: LTSE Phase: Incidence Of Adverse Events Of Special Interest (AESIs)
Description: The primary safety analysis evaluated the effects of OCA treatment on AESIs of pruritus, hepatic disorders, and dyslipidemia. All adverse event (AE) summaries were restricted to treatment emergent AEs (TEAEs), which were defined as any AEs that newly appeared, increased in frequency, or worsened in severity following initiation of investigational product. Treatment-emergent pruritus was defined as any preferred term (PT) including "Prur-". Hepatic disorder AESIs were defined using specific Hepatic Disorders Standardized Medical Dictionary for Regulatory Activities (MedDRA) Query (SMQ) terms. AE lipid profile changes, defined in the Dyslipidemia SMQ, were reported. Verbatim terms were mapped to PTs and system organ classes (SOCs) using MedDRA version 17.1 for all AE summaries except those for hepatic disorder AESIs, which used MedDRA version 18.1. A summary of serious and all other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: LTSE Baseline (DB Week 24) to Month 26
Population: LTSE Population: All participants who received any amount of investigational product during the LTSE phase.
Measure: Count of Participants; unit: Participants
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 59
Participants
  Dyslipidaemia | 1
  Hepatic Disorder | 23
  Pruritus | 34

3. Secondary Outcome: DB Phase: Change From Baseline In Serum Alanine Transaminase (ALT)
Description: As a marker of hepatic biochemistry and liver function, the median change in ALT from Baseline at Week 24 is reported. Results are reported in U/L.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | 1.5 mg OCA Titrating to 3 mg OCA | 5 mg OCA Titrating to 10 mg OCA | Placebo
Number analyzed (Participants) | 25 | 26 | 25
U/L | -33.0 [-50.5 to 5.0] | -5.5 [-30.0 to 4.5] | -19.5 [-49.0 to 4.0]

4. Secondary Outcome: DB Phase: Change From Baseline In Serum Aspartate Aminotransferase (AST)
Description: As a marker of hepatic biochemistry and liver function, the median change in AST from Baseline at Week 24 is reported. Results are reported in U/L.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | 1.5 mg OCA Titrating to 3 mg OCA | 5 mg OCA Titrating to 10 mg OCA | Placebo
Number analyzed (Participants) | 25 | 26 | 25
U/L | -8.0 [-20.0 to 19.0] | 0.5 [-17.5 to 32.8] | -14.0 [-35.5 to 8.0]

5. Secondary Outcome: DB Phase: Change From Baseline In Serum Total Bilirubin
Description: As a marker of hepatic biochemistry and liver function, the median change in serum total bilirubin from Baseline at Week 24 is reported. Results are reported in umol/L.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | 1.5 mg OCA Titrating to 3 mg OCA | 5 mg OCA Titrating to 10 mg OCA | Placebo
Number analyzed (Participants) | 25 | 26 | 25
umol/L | 0.8 [-1.7 to 4.3] | 1.3 [-1.3 to 6.9] | 0.0 [-5.1 to 4.3]

6. Secondary Outcome: DB Phase: Change From Baseline In Serum Direct Bilirubin
Description: As a marker of hepatic biochemistry and liver function, the median change in serum direct bilirubin from Baseline at Week 24 is reported. Results are reported in umol/L.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | 1.5 mg OCA Titrating to 3 mg OCA | 5 mg OCA Titrating to 10 mg OCA | Placebo
Number analyzed (Participants) | 25 | 26 | 25
umol/L | 0.8 [-0.9 to 0.9] | 0.9 [-0.9 to 6.4] | 0.0 [-1.7 to 4.3]

7. Secondary Outcome: DB Phase: Change From Baseline In Serum Gamma-glutamyl Transferase (GGT)
Description: As a marker of hepatic biochemistry and liver function, the median change in serum GGT from Baseline at Week 24 is reported. Results are reported in U/L.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | 1.5 mg OCA Titrating to 3 mg OCA | 5 mg OCA Titrating to 10 mg OCA | Placebo
Number analyzed (Participants) | 25 | 26 | 25
U/L | -79.0 [-171.0 to -9.7] | -78.5 [-235.5 to 14.0] | -89.0 [-167.0 to 20.0]

8. Secondary Outcome: DB Phase: Change From Baseline In Plasma Fibroblast Growth Factor-19 (FGF-19)
Description: To assess farnesoid X receptor (FXR) activity, the change in FGF-19 from Baseline at Week 24 is reported. Results are reported in picograms/milliliter (pg/mL).
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | 1.5 mg OCA Titrating to 3 mg OCA | 5 mg OCA Titrating to 10 mg OCA | Placebo
Number analyzed (Participants) | 25 | 26 | 25
pg/mL | 32.00 [-16.00 to 110.00] | 147.00 [-6.35 to 714.50] | -19.50 [-79.56 to 28.00]

9. Secondary Outcome: DB Phase: Change From Baseline In Plasma 7α-Hydroxy-4-cholesten-3-one (C4)
Description: To assess FXR activity, the change in plasma C4 from Baseline at Week 24 is reported. Results are reported in nanograms (ng)/mL.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | 1.5 mg OCA Titrating to 3 mg OCA | 5 mg OCA Titrating to 10 mg OCA | Placebo
Number analyzed (Participants) | 25 | 26 | 25
ng/mL | -2.80 [-7.50 to 0.55] | -2.90 [-6.94 to -1.12] | 0.05 [-2.25 to 10.84]

10. Secondary Outcome: LTSE Phase: Change From Baseline In Serum ALP At Month 12
Description: The median change in serum ALP from Baseline to the last available visit is reported. The DB value at Week 24 was used as the Baseline. Results are reported in U/L.
Time Frame: LTSE Baseline (DB Week 24), Month 12
Population: LTSE Population: All participants who received any amount of investigational product during the LTSE phase and had an efficacy assessment at the specified time points.
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 34
U/L | -91.5 [-144.0 to -17.0]

11. Secondary Outcome: LTSE Phase: Change From Baseline In Serum ALT At Month 12
Description: As a marker of hepatic biochemistry and liver function, the median change in ALT from Baseline at Month 12 is reported. The DB value at Week 24 was used as the Baseline. Results are reported in U/L.
Time Frame: LTSE Baseline (DB Week 24), Month 12
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 35
U/L | -37.0 [-60.5 to -7.5]

12. Secondary Outcome: LTSE Phase: Change From Baseline In Serum AST At Month 12
Description: As a marker of hepatic biochemistry and liver function, the median change in AST from Baseline at Month 12 is reported. The DB value at Week 24 was used as the Baseline. Results are reported in U/L.
Time Frame: LTSE Baseline (DB Week 24), Month 12
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 35
U/L | -14.5 [-30.5 to 9.5]

13. Secondary Outcome: LTSE Phase: Change From Baseline In Serum Total Bilirubin At Month 12
Description: As a marker of hepatic biochemistry and liver function, the median change in serum total bilirubin from Baseline at Month 12 is reported. The DB value at Week 24 was used as the Baseline. Results are reported in umol/L.
Time Frame: LTSE Baseline (DB Week 24), Month 12
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 34
umol/L | 0.5 [-1.7 to 5.2]

14. Secondary Outcome: LTSE Phase: Change From Baseline In Serum Direct Bilirubin At Month 12
Description: As a marker of hepatic biochemistry and liver function, the median change in serum direct bilirubin from Baseline at Month 12 is reported. The DB value at Week 24 was used as the Baseline. Results are reported in umol/L.
Time Frame: LTSE Baseline (DB Week 24), Month 12
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 34
umol/L | 0.0 [-1.7 to 1.8]

15. Secondary Outcome: LTSE Phase: Change From Baseline In Serum GGT At Month 12
Description: As a marker of hepatic biochemistry and liver function, the median change in serum GGT from Baseline at Month 12 is reported. The DB value at Week 24 was used as the Baseline. Results are reported in U/L.
Time Frame: LTSE Baseline (DB Week 24), Month 12
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 34
U/L | -120.3 [-238.0 to 39.0]

16. Secondary Outcome: LTSE Phase: Change From Baseline In Albumin At Month 12
Description: As a marker of hepatic biochemistry and liver function, the median change in albumin from Baseline at Month 12 is reported. The DB value at Week 24 was used as the Baseline. Results are reported in grams (g)/L.
Time Frame: LTSE Baseline (DB Week 24), Month 12
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: g/L
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 35
g/L | -0.5 [-3.5 to 1.0]

17. Secondary Outcome: LTSE Phase: Change From Baseline In INR At Month 12
Description: As a marker of hepatic biochemistry and liver function, the median change in INR from Baseline at Month 12 is reported. The DB value at Week 24 was used as the Baseline.
Time Frame: LTSE Baseline (DB Week 24), Month 12
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 35
Ratio | 0.0 [0.0 to 0.1]

18. Secondary Outcome: LTSE Phase: Change From Baseline In Transient Elastography (TE) At Month 12
Description: As a marker of hepatic inflammation and fibrosis, the median change in TE, as a measure of hepatic stiffness, from Baseline at Month 12 is reported. The DB value at Week 24 was used as the Baseline. Results are reported in kilopascal (kPa).
Time Frame: LTSE Baseline (DB Week 24), Month 12
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: kPa
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 29
kPa | 1.8 [-0.8 to 6.0]

19. Secondary Outcome: LTSE Phase: Change From Baseline In Enhanced Liver Fibrosis (ELF) At Month 12
Description: As a marker of hepatic inflammation and fibrosis, the change in ELF score from Baseline at Month 12 is reported. The ELF score and its components (hyaluronic acid [HA]; procollagen-3 N-terminal peptide [P3NP]; tissue inhibitor of metalloproteinase 1 [TIMP-1]) was calculated as follows: 2.278 + 0.851 x ln(HA (ng/mL)) + 0.751 x ln(P3NP (ng/mL)) + 0.394 x ln(TIMP-1 (ng/mL). The DB value at Week 24 was used as the Baseline. An increase in score indicates an improvement/worsening of symptoms.
Time Frame: LTSE Baseline (DB Week 24), Month 12
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 34
Units on a scale | 0.3 [0.0 to 1.0]

20. Secondary Outcome: LTSE Phase: Change From Baseline In Plasma FGF-19 At Month 12
Description: To assess FXR activity, the change in FGF-19 from Baseline at Month 12 is reported. The DB value at Week 24 was used as the Baseline. Results are reported in pg/mL.
Time Frame: LTSE Baseline (DB Week 24), Month 12
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 35
pg/mL | 77.7 [-37.0 to 194.0]

21. Secondary Outcome: LTSE Phase: Change From Baseline In Plasma C4 At Month 12
Description: To assess FXR activity, the change in plasma C4 from Baseline at Month 12 is reported. The DB value at Week 24 was used as the Baseline. Results are reported in ng/mL.
Time Frame: LTSE Baseline (DB Week 24), Month 12
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 35
ng/mL | -3.8 [-8.1 to -0.9]

22. Secondary Outcome: LTSE Phase: Participants Experiencing Ulcerative Colitis Remission At Month 12
Description: To assess inflammatory bowel disease (IBD) activity, the number of participants experiencing ulcerative colitis remission at Month 12 is reported. Remission was defined as a partial Mayo score of ≤2 with no individual sub-score exceeding 1 point.
Time Frame: Month 12
Population: LTSE Population: All participants who received any amount of investigational product during the LTSE phase.
Measure: Number; unit: participants
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 59
participants
  Yes | 16
  No | 0

23. Secondary Outcome: LTSE Phase: Participants Experiencing Crohn's Disease Remission At Month 12
Description: To assess IBD activity, the number of participants experiencing Crohn's Disease remission at Month 12 is reported. Remission was defined as a Crohn's Disease Activity Index score of <150.
Time Frame: Month 12
Population: LTSE Population: All participants who received any amount of investigational product during the LTSE phase.
Measure: Number; unit: participants
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 59
participants
  Yes | 5
  No | 1

24. Secondary Outcome: LTSE Phase: Change From Baseline In Total Bile Acids At Month 12
Description: To assess the effects on bile acids, the median change in total bile acids from Baseline at Month 12 is reported. The DB value at Week 24 was used as the Baseline. Results are reported in umol/L.
Time Frame: Month 12
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 35
umol/L | -1.59 [-8.12 to 6.49]

25. Secondary Outcome: LTSE Phase: Change From Baseline In Pruritus Visual Analogue Scale (VAS) At Month 12
Description: To assess the effects on disease-specific symptoms, the median change in the pruritus VAS score from Baseline at Month 12 is reported. The score is derived from the VAS participant questionnaire, which has the participant draw a line anywhere on a scale that best represents the severity of the itch; the scale ranges from 0 (no itching) to 10 (worst possible itching), in increments of 2. An increase in score represents an increase in severity of symptoms. The DB value at Week 24 was used as the Baseline.
Time Frame: LTSE Baseline (DB Week 24), Month 12
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 37
units on a scale | 1.0 [0.0 to 20.0]

ADVERSE EVENTS:
Time Frame: DB Phase: From informed consent to end of double-blind phase study participation, up to 24 weeks. LTSE Phase: Baseline (DB Week 24) to Month 26.
Description: Adverse events reporting is based on the safety population, where the treatment group was defined by the treatment actually received. One (1) placebo participant actually received 5 mg OCA titrating to 10 mg OCA. All adverse event summaries are based on treatment-emergent adverse events. Verbatim terms were mapped to PTs and SOCs using MedDRA version 17.1 for all AE summaries except those for hepatic disorder AESIs, which used MedDRA version 18.1.
Arm/Group | 1.5 mg OCA Titrating to 3 mg OCA | 5 mg OCA Titrating to 10 mg OCA | Placebo | LTSE OCA Total
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/27 | 0/24 | 0/59
Serious Adverse Events (participants affected / at risk) | 4/25 | 4/27 | 2/24 | 19/59
Other Adverse Events (participants affected / at risk) | 20/25 | 24/27 | 21/24 | 53/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.5 mg OCA Titrating to 3 mg OCA (N=25) | 5 mg OCA Titrating to 10 mg OCA (N=27) | Placebo (N=24) | LTSE OCA Total (N=59)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholangitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon dysplasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pouchitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.5 mg OCA Titrating to 3 mg OCA (N=25) | 5 mg OCA Titrating to 10 mg OCA (N=27) | Placebo (N=24) | LTSE OCA Total (N=59)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (31) | 18 (38) | 11 (17) | 33 (62)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 6 (7) | 3 (3) | 8 (10)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (3) | 4 (5) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (3) | 8 (13)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 2 (2) | 4 (4) | 7 (8)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (2) | 4 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 8 (8)
Abdominal distension (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (2) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 2 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 4 (4)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
Pyrexia (General disorders) | 3 (5) | 4 (4) | 1 (1) | 4 (6)
Fatigue (General disorders) | 1 (2) | 3 (3) | 2 (2) | 4 (5)
Oedema peripheral (General disorders) | 1 (3) | 2 (2) | 0 (0) | 3 (4)
Headache (Nervous system disorders) | 2 (3) | 2 (2) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 3 (3) | 3 (3) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 0 (0) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (5) | 1 (1) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Jaundice (Hepatobiliary disorders) | 2 (2) | 1 (1) | 1 (1) | 5 (5)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1) | 3 (3)
Seasonal allergy (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (6)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (3) | 4 (6)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 3 (5)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (3) | 4 (4)

LIMITATIONS AND CAVEATS:
Due to administrative reasons, the study was terminated by the Sponsor prior to most participants completing LTSE Month 24.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators must wait 18 months after the study ends to publish their results and a multi-center publication must come first. The sponsor has a 45-day review period with the option to extend to an additional 90 days.

DOCUMENTS (2):
  • Study Protocol (2016-03-18): https://cdn.clinicaltrials.gov/large-docs/36/NCT02177136/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT02177136/SAP_001.pdf